CLINICAL TRIAL: NCT03335943
Title: The Efficacy and Safety of CDA-2 for the Treatment of IPSS Lower/Intermediate-risk Myelodysplastic Syndrome Patients: a Multi-centered Prospective Open Study
Brief Title: Myelodysplastic Syndrome--CDA-2 Hematological Improvement National Affirmation Study
Acronym: MD-CHINA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Society of Hematology (Other)
Collaborators: Harbin Institute of Hematology & Oncology (Unknown)
Responsible Party: Principal Investigator, Wu Depei, Professor, Chinese Society of Hematology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDA-2 MDS-2017
Record Dates: First submitted 2017-10-17; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: CDA-2, MDS
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CDA-2 (Cell Differentiation Agent 2) (Experimental): Patients will be given CDA-2 therapy.
  Interventions: Drug: CDA-2 (Cell Differentiation Agent 2)

INTERVENTIONS:
Drug: CDA-2 (Cell Differentiation Agent 2) — CDA-2 will be given intravenously, with 200 ml each day for 14 consecutive days in every four weeks (one cycle). The treatment will be repeated at least for 3 cycles.
  Other Names: Uroacitides (a compound mixed of peptides and organic acids)

SUMMARY:
This Study aims to evaluate the efficacy and safety of CDA-2 in the treatment of International Prognostic Scoring System (IPSS) Lower/Intermediate-risk myelodysplastic syndrome (MDS) in Chinese patients.

DETAILED DESCRIPTION:
Patients with lower/intermediate-risk myelodysplastic syndrome (MDS) have rare therapeutic options other than supportive care. In pilot studies, CDA-2 showed promising results of hematological improvement in these patients.

To date, the optimal regimen for CDA-2 treatment is not well established. The researchers are going to make a multi-centered clinical trial to evaluate the efficacy and safety of CDA-2 in 800 patients with International Prognostic Scoring System(IPSS) Lower/Intermediate-risk myelodysplastic syndrome (MDS).

Eligible patients will be given CDA-2 intravenously, with 200 ml each day for 14 consecutive days in every four weeks (one cycle). The treatment will be repeated at least for 3 cycles. The patients will be followed up to 24 weeks.

The primary endpoint is hematological improvement (HI) at 12 weeks according to IWG criteria. Full blood counts will be done on all patients every week. Change in bone marrow function as measured by changes in bone marrow morphology and cytogenetics will be assessed before and after 3 cycles of the treatment.

The secondary endpoint is the therapy response. Complete remission (CR), partial remission (PR) and response duration, side effects, evaluation of QOL will be evaluated at the end of the treatment in every cycle.

Adverse events of the treatment will be recorded for evaluation of the safety.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of MDS according to World Health Organization (WHO)/French American British (FAB) classification that meets IPSS-R classification of low, or intermediate-1 risk disease.
* Subject is 18 to 85years of age the time of signing the informed consent form (ICF).
* Able to adhere to the study visit schedule and other protocol requirements
* Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2.
* Laboratory test results within these ranges: Serum creatinine </=1.5 mg/dL x Upper limit of the normal (ULN),Blood urine nitrogen (BUN)</=1.5 mg/dL x Upper limit of the normal (ULN),Total bilirubin </=1.5 mg/dL x Upper limit of the normal (ULN),Serum glutamic oxaloacetic transaminase/aspartate transaminase (SGOT/AST) and Serum glutamic pyruvic transaminase/alanine transaminase (SGPT/ALT)</=2 x Upper limit of the normal (ULN).
* No prior intensive combination chemotherapy or dose Azacitidine,Decitabine,and Lenalidomide,etc.
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.

Exclusion Criteria:

* IPSS risk group intermediate-2 or high risk
* breast feeding and pregnant women
* MDS associated with del 5q cytogenetic abnormality
* Patients with history of hepatitis B, C, HIV(+), alcoholic liver disease or evidence of hepatopathy will be excluded.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Hematological Improvement (HI) at 12 Weeks | 12 weeks
  Hematologic improvement (HI) per International Working Group (IWG),HI: hemoglobin increase of >= 1.5 g/dL, platelet increase of >= 30,000/mL (starting with > 20,000/mL), neutrophils increase of >= 100% and > 500/μL.

SECONDARY OUTCOMES:
Response Rate of The Therapy at 12 Weeks | 12 weeks
  IWG 2006 response criteria - CR: bone marrow evaluation shows <= 5% blasts; normal maturation of all cells lines (mCR), peripheral blood evaluation shows hemoglobin >= 11 g/dL, neutrophils >= 1000/mL, platelets >= 100,000/mL, 0% blasts; PR: Same as CR, except blasts decrease >= 50%, still greater than 5% in bone marrow
Red Blood Cell Transfusion Independence (RBC-TI) in 24 weeks | 24 weeks
  Proportion of subjects who are Red blood cell (RBC) transfusion free over any consecutive 84-day period within 24 weeks
Change From Baseline to that of the 24 weeks of Scores of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ C-30) Physical Functioning Scale | 24 weeks
  The EORTC QLQ will be evaluated for each patients at the beginning and end of the study.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma X. Epidemiology of myelodysplastic syndromes. Am J Med. 2012 Jul;125(7 Suppl):S2-5. doi: 10.1016/j.amjmed.2012.04.014. PMID 22735748
- [Background] Fenaux P, Haase D, Sanz GF, Santini V, Buske C; ESMO Guidelines Working Group. Myelodysplastic syndromes: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2014 Sep;25 Suppl 3:iii57-69. doi: 10.1093/annonc/mdu180. Epub 2014 Jul 25. No abstract available. PMID 25185242
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Ma+X.+The+American+journal+of+medicine.+2012%3B125(7+Suppl)%3AS2-5.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Fenaux+P%2C+Haase+D%2C+Sanz+GF%2C+Santini+V%2C+Buske+C%2C+Group+EGW.+Annals+of+oncology+%3A+official+journal+of+the+European+Society+for+Medical+Oncology+%2F+ESMO.